CLINICAL TRIAL: NCT03538678
Title: Just Kwit: Mobile Intervention for Tobacco Cessation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Kar-Hai Chu, Assistant Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: PRO18010454; K07CA222338 (NIH)
Record Dates: First submitted 2018-04-14; First posted 2018-05-29 (Actual); Results first posted 2021-02-18 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kwit app (Experimental): Use of Kwit smartphone app
  Interventions: Other: Kwit smartphone app
- Standard of care (No Intervention): Patient initiated follow-up post discharge

INTERVENTIONS:
Other: Kwit smartphone app — Kwit smarphone app
  Arms: Kwit app

SUMMARY:
The intervention will be use of a smartphone app to support tobacco cessation. The app's main features include sending motivational messages, displaying money saved, and allowing the user to log cravings.

DETAILED DESCRIPTION:
The investigators will recruit hospitalized young adult smokers aged 18-30 interested in cessation over a six-month period. Patients will all receive a UPMC Tobacco Treatment Service counseling session focused on motivational interviewing prior to participation in the study. Upon consent, participants will then be randomized 1:1 to either standard patient-initiated follow-up or use of the Kwit app. Participants will be stratified by sex because males and females are known to have highly variable responses to existing tobacco control interventions. Investigators will systematically assess feasibility using established Likert-type items factors such as interaction, features, engagement, trust, and impact.

If a participant consents to the study, they will be given a brief survey to collect general information related to their smoking behavior. After 30 days, a follow-up survey will be conducted to assess their current smoking behavior. Participants randomized to the experimental arm will be asked additional questions about their use of the smartphone app.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-30 smokers interested in cessation (>5 cigarettes/day over the past 30 days)
* Must own an Apple or Android based smartphone.

Exclusion Criteria:

* Already receiving pharmacological and/or behavioral intervention or counseling for smoking cessation.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2018-06-11 (Actual); Primary Completion 2019-12-29 (Actual); Study Completion 2019-12-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kar-Hai Chu, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chu KH, Escobar-Viera CG, Matheny SJ, Davis EM, Primack BA. Tobacco cessation mobile app intervention (Just Kwit! study): protocol for a pilot randomized controlled pragmatic trial. Trials. 2019 Feb 26;20(1):147. doi: 10.1186/s13063-019-3246-2. PMID 30808389

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Kwit App | Standard of Care
Started | 20 | 20
Completed | 5 | 9
Not Completed | 15 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Kwit App | Standard of Care | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Customized [Count of Participants; unit: Participants]
  <18 | 0 | 0 | 0
  >=18 and <=30 | 20 | 20 | 40
  >30 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 10 | 10 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 20 | 20 | 40
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 3 | 8
  White | 13 | 16 | 29
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Feasibility - Helpfulness and Ease of Use of the Intervention Smartphone App
Description: Assessment of feasibility - Descriptive statistics that will be obtained via a follow up survey will be used to assess feasibility. The follow up survey will be administered one month after discharge via email, phone or in-person, determined by the preference of the participant. Specific questions will be asked asking participants to rate the Kwit smartphone application based on helpfulness, ease of use, and to list frustrations and helpful aspects of the application.
  How helpful was the Kwit app? Very helpful Somewhat helpful Neutral Not very helpful Not at all helpful
  Was the app easy to use? Very Somewhat Neutral Not much Not at all
  Was it frustrating to use? Very Somewhat Neutral Not much Not at all
  What, if anything, was helpful about the app? What, if anything, was not helpful about the app?
Time Frame: 1-month
Population: Only applicable for experimental arm
Measure: Count of Participants; unit: Participants
Arm/Group | Kwit App | Standard of Care
Number analyzed (Participants) | 5 | 0
Participants
  App helpful: Very | 2 |
  App helpful: Somewhat | 2 |
  App helpful: Neutral | 1 |
  App helpful: Not very | 0 |
  App helpful: Not at all | 0 |
  App easy to use: Very | 3 |
  App easy to use: Somewhat | 2 |
  App easy to use: Neutral | 0 |
  App easy to use: Not very | 0 |
  App easy to use: Not at all | 0 |
  App frustrating to use: Very | 0 |
  App frustrating to use: Somewhat | 1 |
  App frustrating to use: Neutral | 0 |
  App frustrating to use: Not very | 2 |
  App frustrating to use: Not at all | 2 |

2. Primary Outcome: Feasibility - Frequency of Use
Description: Assessment of feasibility - Descriptive statistics that will be obtained via a follow up survey will be used to assess feasibility. The follow up survey will be administered one month after discharge via email, phone or in-person, determined by the preference of the participant. Specific questions will be asked asking participants to rate the Kwit smartphone application based on frequency of use.
Time Frame: 1-month
Population: Only applicable for experimental arm
Measure: Count of Participants; unit: Participants
Arm/Group | Kwit App | Standard of Care
Number analyzed (Participants) | 5 | 0
Participants
  Almost everyday | 0 |
  Several days/week | 2 |
  Several days/month | 3 |
  Not at all | 0 |

3. Secondary Outcome: Cessation--point Prevalence Abstinence
Description: Assessment of cessation - Descriptive statistics will be used to assess cessation outcomes. The information will be obtained via a follow up survey with specific questions pertaining to the level of participant smoking as well as their confidence levels on maintaining cessation.
  Since you left the hospital in (month/year), have you smoked a cigarette (even a puff)?
  In the past 30 days, have you smoked a cigarette, even a puff?
  In the past 7 days, have you smoked a cigarette, even a puff?
Time Frame: 1-month
Measure: Count of Participants; unit: Participants
Arm/Group | Kwit App | Standard of Care
Number analyzed (Participants) | 5 | 9
Participants
  Smoke since leaving hospital: Yes | 4 | 8
  Smoke since leaving hospital: No | 1 | 1
  Smoke since leaving hospital: Don't know | 0 | 0
  Smoke since leaving hospital: Did not answer | 0 | 0
  Smoke past 30 days: Yes | 3 | 8
  Smoke past 30 days: No | 0 | 0
  Smoke past 30 days: Don't know | 1 | 0
  Smoke past 30 days: Did not answer | 1 | 1
  Smoke past 7 days: Yes | 4 | 5
  Smoke past 7 days: No | 0 | 3
  Smoke past 7 days: Don't know | 0 | 0
  Smoke past 7 days: Did not answer | 1 | 1

4. Secondary Outcome: Cessation--cigarettes Smoked
Description: Assessment of cessation - Descriptive statistics will be used to assess cessation outcomes. The information will be obtained via a follow up survey with specific questions pertaining to the level of participant smoking as well as their confidence levels on maintaining cessation.
  (On the days you smoked), how many cigarettes on average did you smoke (even a puff)?
Time Frame: 1-month
Population: 4 participants (2 exp, 2 control) did not answer this question.
Measure: Mean (Standard Deviation); unit: Cigarettes smoked
Arm/Group | Kwit App | Standard of Care
Number analyzed (Participants) | 3 | 7
Cigarettes smoked | 4.67 (0.58) | 8.14 (5.49)

5. Secondary Outcome: Cessation--days Smoked
Description: Assessment of cessation - Descriptive statistics will be used to assess cessation outcomes. The information will be obtained via a follow up survey with specific questions pertaining to the level of participant smoking as well as their confidence levels on maintaining cessation.
  In the past 30 days, on how many days did you smoke (even a puff)?
Time Frame: 1-month
Population: 5 participants (2 exp, 3 control) did not answer this question.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Kwit App | Standard of Care
Number analyzed (Participants) | 3 | 6
Days | 21.67 (7.64) | 17.67 (12.97)

6. Secondary Outcome: Cessation--confidence
Description: Assessment of cessation - Descriptive statistics will be used to assess cessation outcomes. The information will be obtained via a follow up survey with specific questions pertaining to the level of participant smoking as well as their confidence levels on maintaining cessation.
  How confident are you that you will be able to stay quit?
Time Frame: 1-month
Population: 2 participants (1 exp, 1 control) did not answer this question.
Measure: Count of Participants; unit: Participants
Arm/Group | Kwit App | Standard of Care
Number analyzed (Participants) | 4 | 8
Participants
  Not at all confident | 1 | 1
  A little confident | 0 | 0
  Somewhat confident | 1 | 3
  Fairly confident | 1 | 2
  Very confident | 1 | 1
  Don't know | 0 | 0
  Refuse to answer | 0 | 0
  N/A | 0 | 1

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | Kwit App | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

LIMITATIONS AND CAVEATS:
Primary purpose of trial was to study feasibility, with limited analyses planned. With low follow-up, statistical analyses would not be appropriate.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2019-06-06): https://cdn.clinicaltrials.gov/large-docs/78/NCT03538678/Prot_000.pdf